CLINICAL TRIAL: NCT01238081
Title: The Role of Respiratory Viruses in Exacerbations of Cystic Fibrosis in Adults.
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2010CF004
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Respiratory viruses, such as those that cause colds and influenza, are very common in the general population. The average adult will experience between 2 and 4 viral respiratory illnesses each year. It is known that respiratory viruses can cause flare-ups of chronic lung diseases such as asthma and chronic obstructive pulmonary disease. In children with CF, respiratory viral infections have been identified in nearly half of all exacerbations and are associated with a decline in lung function and increased frequency of hospital admission and acquisition of new bacterial pathogens.

Currently, little is known about the impact of viral infections on the course of CF lung disease in adults and no large-scale prospective studies in this area have been performed to date. It is unknown how often respiratory viruses can be found in patients with CF when they are well and what consequences they have on the course of exacerbations of CF lung disease. This study will identify the frequency of common viral infections in adults with CF and determine the effects they have on lung function, the rate and diversity of bacterial infection and patients' treatment burden. The information gained from this study will lead to improved prevention and treatment of respiratory infections in CF.

DETAILED DESCRIPTION:
Background Lung disease in cystic fibrosis (CF) is characterized by chronic airway infection with periodic exacerbations which are associated with impaired lung function, reduced quality of life and increased healthcare costs.1 2 Respiratory viruses are common and are known to be associated with exacerbations of other chronic respiratory diseases such as asthma.3 Studies in children with CF have shown that respiratory viruses are common during exacerbations. Wat and colleages identified respiratory viruses in 46% of patients at the time of pulmonary exacerbation of CF.4 Several older studies in children with CF have found an association between viral infections and decline in lung function, frequency and duration of hospital admission and CF disease progression.5-7 An association between respiratory viruses and acquisition of Pseudomonas aeruginosa has been proposed but this remains unproven.8 Retrospective data in adults has shown an incidence of viral infection in pulmonary exacerbations of between 8.7 and 45.8%.9 10 To date, no prospective studies have been conducted to investigate the impact of these infections on clinical outcomes in adults with CF, or the effects of these infections on respiratory bacterial flora. It is entirely unknown how frequently viruses can be identified in adults with CF when they are asymptomatic. This study will fill these gaps in current knowledge and improve our management of respiratory infections in CF.

Primary Research Question What is the prevalence of respiratory virus infection in adults with CF during a pulmonary exacerbation and when clinically stable?

Secondary Research Questions

1. What is the effect of respiratory virus infection on lung function and disease progression?
2. What is the effect of respiratory virus infection on bacterial and fungal colonization in CF?
3. What is the effect of respiratory virus infection on the CF microbiome, specifically the rate and diversity of bacterial infection?
4. Are any specific rhinovirus sub-types (including rhinovirus C) associated with worse outcome following viral respiratory infections in adults with CF?

Methodology This is a prospective observational study looking at the incidence and consequences of respiratory virus infection in CF both during exacerbations and during periods of clinical stability. Subjects eligible for the study will be all patients with CF over the age of 18 years attending the Manchester Adult Cystic Fibrosis Centre (MACFC). We aim to recruit 100 patients into the study. Participants will be screened for respiratory viruses at baseline and every two months throughout a twelve month follow-up period. Screening will also occur at the time of diagnosis of a pulmonary exacerbation or onset of new respiratory symptoms. At each visit an oral mouth wash, sputum sample and a nose-swab will be taken; the mouth wash and an aliquot of sputum will be stored frozen for later microbial diversity analysis. On each occasion, sputum will also be sent for conventional bacteriology/mycology to identify any new bacterial or fungal colonization.

Respiratory viruses in the sputum will then be identified using the polymerase chain reaction (PCR) technique. The following viruses will be tested for: adenovirus, human metapneumovirus, influenza A, B & C (including influenza A H1N1), parainfluenza 1-3, respiratory syncytial virus and rhinovirus. Rhinovirus identifications will be sequenced to determine the frequency of infection with individual subtypes.

After 6 months of the study, 10 CF individuals who provided a stable and viral-linked exacerbation samples will be selected and the total bacterial diversity in their sputum examined by state-of-the-art, cultivation independent 16S rRNA pyrosequencing analysis.11 To account for the potential of oral flora contamination in the sputum samples, the mouth wash taken prior to each sputum sample will also be examined. Total DNA will be extracted from the selected samples and the V1-3 region of the 16S rRNA gene amplified using tagged primers specifically developed for pyrosequencing sequence analysis. The derived bacterial 16S rRNA gene sequences (8000-10,000 reads per sample) will be trimmed to 450 bases and compared to the Ribosomal Database Project (RDP; http://rdp.cme.msu.edu) to determine the identity of the bacteria from which the DNA derived. Correlation between viral-linked exacerbation and the load of known pathogens (eg. Pseudomonas aeruginosa), new players (CF anaerobes), and the total/unique bacterial flora in the sputum will be made.

Data Analysis & Statistical Methods The primary outcome measure will be identification of a respiratory virus in nose/throat swab or sputum. Statistical analysis will use longitudinal regression modeling of the cohort which takes account of the repeated sampling of each patient. The study will have over 80% power to detect differences of 20% (e.g. 50% vs. 30%) in incidence of viral infection between exacerbation and routine sample periods in patients showing at least one-third of the samples with infection (using a McNemar's paired test with p=0.05).

Ethical Approval The study has been reviewed by the North West 9 Research Ethics Committee - Greater Manchester West and has received a favourable opinion.

References

1. Goss C et al. Exacerbations in cystic fibrosis. 1: Epidemiology and pathogenesis. Thorax 2007;62:360-7.
2. Britto M et al. Impact of recent pulmonary exacerbations on quality of life in patients with cystic fibrosis. Chest 2002;121:64-72.
3. Johnston S et al. The relationship between upper respiratory infections and hospital admissions for asthma: a time-trend analysis. Am J Respir Crit Care Med 1996;154:654-60.
4. Wat D et al. The role of respiratory viruses in cystic fibrosis. J Cystic Fibros 2008;7:320-8.
5. Smyth A et al. Effect of respiratory virus infections including rhinovirus on clinical status in cystic fibrosis. Arch Dis Child 1995;73:117-20.
6. Wang E et al. Association of respiratory viral infections with pulmonary deterioration in patients with cystic fibrosis. N Engl J Med 1984;311:1653-8.
7. Collinson J et al. Effects of upper respiratory tract infections in patients with cystic fibrosis. Thorax 1996;51:1115-22.
8. Petersen NT et al. Respiratory infections in cystic fibrosis patients caused by virus, chlamydia and mycoplasma--possible synergism with Pseudomonas aeruginosa. Acta Paed Scand 1981;70:623-8.
9. De Schutter I et al. Detection of viruses in pulmonary exacerbations in CF. J Cystic Fibros, 2010:s37.
10. Naseer R et al. Pulmonary exacerbations in adult patients with cystic fibrosis associated with positive viral PCR. J Cystic Fibros 2010;9:S37.

11 White J et al. Culture-independent analysis of bacterial fuel contamination provides insights into the level of concordance with conventional cultivation. Appl Environ Microbiol (in review) 2010.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cystic fibrosis attending Manchester Adult CF Centre
* Age ≥18 years
* Capable of providing written informed consent
* Able and willing to provide required samples and meet visit schedule

Exclusion Criteria:

* Previous lung transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with cystic fibrosis attending the Manchester Adult Cystic Fibrosis Centre, Manchester, UK
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Identification of respiratory viruses in sputum, nose- or throat-swabs | 12 months
  A panel of 6 viruses will be tested for using polymerase chain reaction (PCR)technology: adenovirus, rhinovirus, metapneumovirus, parainfluenza virus 1-3, influenza A,B&C and respiratory syncytial virus

CONTACTS AND LOCATIONS:
Overall Officials: William G Flight, MBChB, Principal Investigator — University Hospital of South Manchester NHS FoundationTrust
Locations (1):
- University Hospital of South Manchester NHS Foundation Trust, Manchester, Lancashire, United Kingdom

REFERENCES:
- See also: UK Cystic Fibrosis Trust — http://www.cftrust.org.uk
- See also: University Hospital of South Manchester — http://www.uhsm.nhs.uk